CLINICAL TRIAL: NCT06536218
Title: Effects of Mindfulness Stress Reduction Program on Sleep Status, Stress and Quality of Life in Patients With Sleep Disorders: A Polysomnographic Study
Brief Title: Sleep Disorder Mindfulness Stress Reduction Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MAUN
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Patients in the Sleep Clinic
Keywords: SLEEPING DISORDER; POLYSOMNOGRAPHIC RESEARCH; CONSCIOUS AWARENESS; LIFE QUALITY; STRESS

STUDY DESIGN:
Intervention Model Description: Conscious awareness is a skill that is inherent in human nature and can be developed through training and programs. This skill will provide the individual with the opportunity to achieve inner peace, help him find ways to cope with stress and make him feel less anxiety. Internalization of the skills gained by doing conscious awareness practices is related to the participation of the individuals in the group in the process and their individual experiences in performing the practices. Although group support is effective in the acquisition of these skills, using the acquired skills in daily life is also important for the continuity of the level of conscious awareness (Mason and Hargreaves, 2001).
Masking Description: Control Group; It is planned to conduct a one-session (60-minute), unstructured, active participation-based group application (the week when the first session is applied to the intervention group) in which participants share their experiences with each other about stress and stressful experiences.
  Intervention Group: Conscious Awareness Based Stress Reduction (BFTSA) intervention consists of seven sessions in total and is planned to be completed in a total of seven weeks, with one session per week and each session being 45 minutes. After the results of the patients who underwent PSG are determined according to the randomization criteria and receive certain points from the sleep scale, it is planned to call the patients by phone and explain the meaning and importance of the study, the applications to be performed in the study and its duration. It is planned to have an online individual interview with patients who agree to participate in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): It is planned to conduct a one-session (60-minute), unstructured, active participation-based group application (the week when the first session is applied to the intervention group) in which participants share their experiences with each other about stress and stressful experiences.
- CONSCIOUS AWARENESS STRESS REDUCTION PROGRAM APPLICATION (Experimental): Conscious Awareness Based Stress Reduction (BFTSA) intervention consists of seven sessions in total and is planned to be completed in a total of seven weeks, with one session per week and each session being 45 minutes. After the results of the patients who underwent PSG are determined according to the randomization criteria and receive certain points from the sleep scale, it is planned to call the patients by phone and explain the meaning and importance of the study, the applications to be performed in the study and its duration. It is planned to have an online individual interview with patients who agree to participate in this study.
  Interventions: Behavioral: CONSCIOUS AWARENESS STRESS REDUCTION PROGRAM APPLICATION

INTERVENTIONS:
Behavioral: CONSCIOUS AWARENESS STRESS REDUCTION PROGRAM APPLICATION — CONSCIOUS AWARENESS STRESS REDUCTION PROGRAM APPLICATION Conscious Awareness Based Stress Reduction (BFTSA) intervention consists of seven sessions in total and is planned to be completed in a total of seven weeks, with one session per week and each session being 45 minutes. After the results of the PSG patients are determined according to the randomization criteria, they receive certain points from the sleep scale, it is planned to call the patients by phone and explain the meaning and importance of the study, the applications to be performed in the study and its duration. It is planned to hold online individual interviews with patients who agree to participate in this study.
  Arms: CONSCIOUS AWARENESS STRESS REDUCTION PROGRAM APPLICATION

SUMMARY:
Sleep problems, ranging from mild sleep disturbance to debilitating insomnia, are among the most common health problems occurring in adults, with an estimated prevalence of 35% to 48% (Morin et al., 2009; Mai and Buyss 2008). Insomnia is a fairly common sleep disorder characterized by difficulty falling asleep, difficulty staying asleep, or waking up too early despite adequate sleep opportunity, recurring at least three times a week and accompanied by significant stress or distress during the day (Morin and Jarrin, 2013). ). According to the American guidelines for the treatment of chronic insomnia published in 2017, pharmacotherapy and non-pharmacological treatment are the two main treatment methods for sleep disorders ( Sateia et al., 2017 ).Mindfulness-based stress reduction (MBSR) is an important type of non-pharmacological mindfulness-based intervention that effectively relieves insomnia by decentering (Banno et al., 2019).Regarding the effect of mindfulness intervention in sleep disorders, Ong and Moore suggest that mindfulness can improve sleep by reducing both primary and secondary arousal (Ong and Moore, 2020).Therefore, this study aims to expand the existing investigations by examining whether mindfulness meditation (MBSR) is associated with changes in objectively measured polysomnographic (PSG) sleep profiles of patients with sleep disorders who applied to the Sleep EMG department of Muş State Hospital, and to examine the changes in PSG sleep in the context of a randomized controlled trial. It aims to determine the effect on quality of life by associating it with subjectively reported sleep and stress changes.

DETAILED DESCRIPTION:
Sleep problems, ranging from mild sleep disturbance to debilitating insomnia, are among the most common health problems occurring in adults, with an estimated prevalence of 35% to 48% (Morin et al., 2009; Mai and Buyss 2008). Insomnia is a fairly common sleep disorder characterized by difficulty falling asleep, difficulty staying asleep, or waking up too early despite adequate sleep opportunity, recurring at least three times a week and accompanied by significant stress or distress during the day (Morin and Jarrin, 2013). ). According to the American guidelines for the treatment of chronic insomnia published in 2017, pharmacotherapy and non-pharmacological treatment are the two main treatment methods for sleep disorders ( Sateia et al., 2017 ).Mindfulness-based stress reduction (MBSR) is an important type of non-pharmacological mindfulness-based intervention that effectively relieves insomnia by decentering (Banno et al., 2019).Regarding the effect of mindfulness intervention in sleep disorders, Ong and Moore suggest that mindfulness can improve sleep by reducing both primary and secondary arousal (Ong and Moore, 2020).A limited but growing body of evidence suggests that mindfulness and other types of meditation may improve sleep quality. Neuondorf et al., (2015) reviewed 112 research studies of insomnia or sleep disturbance testing a variety of different mind-body interventions, including meditation, and found that although the evidence was heterogeneous, limited, and potentially biased, mind-body training was a treatment option for patients. It has been shown that it can be accepted as (Neuendorf et al., 2015). A recent systematic review and meta-analysis focused on identifying and evaluating the clinical significance of different mindfulness-based interventions (MBI) on sleep in individuals with anxiety and depression, showing significant effects on sleep problem improvement across all MBI programs (Chan et al. al., 2022) .Therefore, this study aims to expand the existing investigations by examining whether mindfulness meditation (MBSR) is associated with changes in objectively measured polysomnographic (PSG) sleep profiles of patients with sleep disorders who applied to the Sleep EMG department of Muş State Hospital, and to examine the changes in PSG sleep in the context of a randomized controlled trial. It aims to determine the effect on quality of life by associating it with subjectively reported sleep and stress changes.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65

  * Knowing how to read and write
  * Being able to speak Turkish fluently
  * Being diagnosed with a sleep disorder as a result of Polysomnography

Exclusion Criteria:

* • Being diagnosed with any mental illness

  * Using any psychotropic medication
  * Having a chronic disease that prevents you from doing exercises
  * Participating in any awareness-based training program in the last year
  * Being diagnosed with obstructive sleep apnea syndrome (OSAS)
  * Being diagnosed with narcolepsy

Randomization Criteria In this study, individuals;

* Age,
* Gender,
* Sleep quality scale score,
* Perceived Stress Scale score
* Will be randomized according to quality of life scale scores.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Status | 11 WEEKS
  Conscious Awareness Stress Reduction Program does not affect the sleep status of patients with sleep disorders.
Perceived Stress | 11 WEEKS
  Mindfulness Stress Reduction Program Affects the perceived stress level of patients with sleep disorders
Life quality | 11 WEEKS
  Conscious Awareness Stress Reduction Program affects the quality of life of patients with sleep disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No